CLINICAL TRIAL: NCT06040853
Title: Evaluation of Postoperative Pain in Laparoscopic Radical Prostatectomy Surgery With Tranexamic Acid: Analgesia? Hiperalgesia?
Brief Title: Postoperative Pain in Laparoscopic Radical Prostatectomy Surgery With Tranexamic Acid: Analgesia? Hiperalgesia?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nihan Yaman Mammadov, MD, principal investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: traneksamicanalgesia
Record Dates: First submitted 2023-04-17; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Pharmacological Action
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tranexamic group (Experimental): After intubation, intravenous 15mg/kg tranexamic acid will be given to the study group 10 minutes before the incision and 100 mg/h infusion will be administered until the skin is closed.
  Interventions: Drug: Tranexamic acid intravenous administration
- placebo group (Placebo Comparator): The control group will be given intravenous 100 ml of saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tranexamic acid intravenous administration — Participants will be given 15mg/kg tranexamic acid before the incision in ten minutes, 100 mg/h will continue until the end of the surgery.
  Other Names: intravenous saline administration
  Arms: tranexamic group
Drug: Saline — Participant was given intravenous 100 ml saline
  Other Names: intravenous saline administration
  Arms: placebo group

SUMMARY:
Prostate cancer is the most diagnosed cancer among men today. Radical prostatectomy is a surgery that significantly reduces disease-related mortality. The laparoscopic technique, on the other hand, is preferred because it shortens the hospital stay, faster recovery and less postoperative pain.In this study, it was planned to investigate the analgesic or hyperalgesic effects of tranexamic acid, which is widely used in the management of bleeding in trauma, orthopedic, genitourinary and gynecological surgeries. Routine noninvasive monitoring (ECG, Spo2, NIBP) will be performed when participatient are taken to the operating table without premedication. After midazolam is administered, intubation will be performed by administering 1mg/kg lidocaine, 3mg/kg propofol, 2mcg/kg fentanyl, 0.6mg/kg rocuronium. Anesthesia will be maintained with desflurane with a MAC of 1. A 0.1-0.5 mcg/kg/min remifentanil infusion will be administered by targeting 40-60 values with BIS monitoring. After intubation, 15mg/kg tranexamic acid will be given 10 minutes before the incision, and 100 mg/h infusion will be administered until the skin is closed. The control group will be given 100 ml of saline.1mg/kg tramadol and 1gr parol will be administered 30 minutes before the end of the operation. The primary objectives of the study were to learn the VAS (Visual analog scale) score at 0.6,12, 24,48,72 hours, time to first analgesic requirement, and analgesic requirement within 24 hours. Secondary purposes are to determine the amount of antiemetic used, at the beginning of the operation, Hg at the first hour and postoperative 6 hours, complications and side effects (such as DVT, pulmonary embolism).

DETAILED DESCRIPTION:
Prostate cancer is the most diagnosed cancer among men today. Radical prostatectomy is a surgery that significantly reduces disease-related mortality. The laparoscopic technique, on the other hand, is preferred because it shortens the hospital stay, faster recovery and less postoperative pain.In this study, it was planned to investigate the analgesic or hyperalgesic effects of tranexamic acid, which is widely used in the management of bleeding in trauma, orthopedic, genitourinary and gynecological surgeries

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic radical prostatectomy will be performed; Surgeon with more than 10 years of laparoscopic prostatectomy experience
* Participant BMI(weight/height2)(kg/m2)<35
* ASA2-3
* Participant Age>18
* Participant Age<75

Exclusion Criteria:

* Coagulation disorder,
* Chronic renal failure,
* Patients allergic to tranexamic acid,
* Participant Age<18
* Participant Age>75,
* Participant BMI(weight/height2)(kg/m2)>35,
* Surgeon with less than 10 years of laparoscopic prostatectomy experience,
* Patients who had a cerebral, coronary and thromboembolic event within 6 months before the operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale, time of first analgesic requirement, used within 24 hours amount of analgesic, | Change from baseline at 0., 6., 12., 24., 48., 72. hours VAS score
  Investigators will evaluate VAS score, time of first analgesic requirement, used within 24 hours amount of analgesic,

SECONDARY OUTCOMES:
side effect, 0., 1., 6. hours hemogram value, amount of antiemetic used | Change from baseline at 0., 1., 6. hours
  Investigators will evaluate demographic characteristics [years, female/male, weight(kg),height(meter), BMI (kg/m2 )], side effect, 0,1,6 st hour hemogram value, amount of antiemetic used.

CONTACTS AND LOCATIONS:
Overall Officials: Gülten Arslan, Study Director — DrLutfiKirdar training and research hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arslan G, Mammadov NY, Onal C, Mavi F, Geyik FD, Eler Cevik B. Postoperative pain evaluation in laparoscopic radical prostatectomy surgery using tranexamic acid: analgesia?, hyperalgesia?? World J Urol. 2025 May 13;43(1):300. doi: 10.1007/s00345-025-05581-w. PMID 40358732
- Available data/document: Study Protocol: doi: 10.1371 — https://pubmed.ncbi.nlm.nih.gov/28282425/